CLINICAL TRIAL: NCT03257683
Title: RANOLAZINE STUDY: The Effect of Ranolazine on Speckle Tracking Derived Myocardial Strain in Regions of Non-Revascularizable Ischemic Myocardium
Brief Title: RANOLAZINE STUDY: Speckle Tracking Derived Myocardial Strain
Status: Withdrawn | Type: Observational
Why Stopped: Lack of funding
Sponsor: Saint Thomas Health (Other)
Responsible Party: Sponsor
Other Study IDs: STH 16-012
Record Dates: First submitted 2017-07-25; First posted 2017-08-22 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Severe Coronary Artery Disease; Ischaemic Myocardial Dysfunction
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ranolazine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Selected group with cardiac ischemia: This selected study group will have a specific echocardiographic imaging protocol performed, which includes the known ischemic regions. All segments will be collected and analyzed as a pre-therapeutic baseline using specialized STE software to derive strain values. Following eight (8) weeks of ranolazine therapy, each subject will be re-interrogated with the same echocardiographic imaging protocol and have identical measurements of regional strain performed. Ranolazine will be added to the patients' usual medical therapy. Each patient will serve as their own control, from baseline to post therapeutic state.
  Interventions: Drug: Ranolazine

INTERVENTIONS:
Drug: Ranolazine — Study group will receive additional therapeutic dosing of drug.

SUMMARY:
The purpose of this study is to collect data to determine if the medication, Ranolazine, effects heart muscle function in patients who have areas of non-revascularizable heart muscle.

DETAILED DESCRIPTION:
Many cardiac patients with severe coronary artery disease have areas of ischemic LV myocardium that cannot be revascularized (Non-R). The investigators propose to identify such patients via retrospective case review of CMRI data, as well as identify the exact regions which specify Non-R coronary anatomy. This selected study group will have a specific echocardiographic imaging protocol performed, which includes the known ischemic regions. All segments will be collected and analyzed as a pre-therapeutic baseline using specialized STE software to derive strain values. Following eight (8) weeks of ranolazine therapy, each subject will be re-interrogated with the same echocardiographic imaging protocol and have identical measurements of regional strain performed. Ranolazine will be added to the patients' usual medical therapy. Each patient will serve as their own control, from baseline to post therapeutic state.

It is the hypothesis of the investigators, that additional therapeutic dosing of ranolazine will improve regional and perhaps global myocardial function. Improvement in LV mechanical function (regional and global) will be quantitated and objectively elucidated by STE derived myocardial strain as described further in this document.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 Stable GDMT for 60 days prior to enrollment Normal sinus rhythm Coronary artery revascularization > 60 days prior to enrollment Non-revascularizable area of myocardial ischemia as determined by stress MRI Able to perform the bicycle stress echocardiograms Able to provide written, informed consent Women of childbearing potential with negative pregnancy test at the index visit, and consent to use effective contraception throughout the study period and up to at least 14 days following the last dose of study drug

Exclusion Criteria:

* More than 1+MR, aortic stenosis, aortic insufficiency, mitral stenosis Serious co-morbidities with predicted life expectancy <1 year Patients not in normal sinus rhythm (NSR) Patients who have undergone coronary artery revascularization (PCI, CABG) within 60 days Pregnant or unknown pregnancy status Liver cirrhosis Patients unwilling/unable to provide written, informed consent Concomitant use of QTc prolonging drugs, potassium channel variants resulting in a long QT interval, patients with a family history of (or congenital) long QT syndrome, and patients with known acquired QT interval prolongation Concomitant use of strong CYP3A inhibitors including ketoconazole, itraconazole, clarithromycin, nefazodone, nelfinavir, ritonavir, indinavir, and saquinavir Concomitant use of CYP3A4 inducers such as rifampin, rifabutin, rifapentine, phenobarbital, phenytoin, carbamazepine, and St. John's wort Breast feeding Atrial fibrillation or frequent atrial or ventricular ectopy Moderate CYP3A inhibitors (e.g., diltiazem, verapamil, erythromycin) P-gp inhibitors (e.g., cyclosporine) which increase ranolazine exposure Renal failure. Patients with Creatinine clearance less than 30ml/min . Safety Considerations for patients with the following drugs/conditions CYP3A substrates: Limit simvastatin to 20 mg when used with ranolazine. Doses of other sensitive CYP3A substrates (e.g., lovastatin) and CYP3A substrates with narrow therapeutic range (e.g., cyclosporine, tacrolimus, sirolimus) may need to be reduced with ranolazine OCT2 substrates: Limit the dose of metformin to 1700 mg daily when used with ranolazine 1000 mg twice daily. Doses of other OCT2 substrates may require adjusted doses Drugs transported by P-gp (e.g., digoxin), or drugs metabolized by CYP2D6 (e.g., tricyclic antidepressants) may need reduced doses when used with ranolazine Renal failure: Patients with creatinine clearance less than 30ml/min are excluded from participation in this study. Monitor renal function after initiation and periodically in patients with moderate to severe renal impairment (CrCL < 60 mL/min). If acute renal failure develops, discontinue ranolazine.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will be either male or female, age 18 or greater with stable GDMT for 60 days prior to enrollment. They will be in normal sinus rhythm with coronary artery revascularization more than 60 days prior to enrollment, with a non-revascularizable area of myocardial ischemia as determined by stress MRI. They will be able to perform the bicycle stress echocardiogram and able to provide written informed consent.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-04-14 (Actual); Primary Completion 2017-11-16 (Actual); Study Completion 2018-02-16 (Actual)

PRIMARY OUTCOMES:
Measurement of strain | 8 weeks
  Changes in 3D regional left ventricular myocardial strain assessed by speckle-tracking

SECONDARY OUTCOMES:
Left ventricular function | 8 weeks
  2D global longitudinal strain and various other echo parameters of left ventricular function

CONTACTS AND LOCATIONS:
Overall Officials: Douglas J Pearce, MD, Principal Investigator — Saint Thomas Health
Locations (1):
- Saint Thomas Heart at Saint Thomas West, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No